CLINICAL TRIAL: NCT05072119
Title: Registry of Patients Underwent Cardiac Implanted Electronic Device Implantation at Monaldi Hospital
Brief Title: Monaldi Hospital Rhythm Registry
Status: Recruiting | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Vincenzo Russo, Principal Investigator, University of Campania Luigi Vanvitelli
Other Study IDs: 22052021
Record Dates: First submitted 2021-09-14; First posted 2021-10-08 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Pacemaker; ICD; Implanted Loop Recorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with PM: All patients underwent PM implantation
  Interventions: Device: Device implantation
- Patients with ICD: All patients undeerwent ICD implantation
  Interventions: Device: Device implantation
- Patients with ILR: All patients underwent ILR implantation
  Interventions: Device: Device implantation

INTERVENTIONS:
Device: Device implantation — Implantation of single chamber, dual chambers or triple chambers PM/ICD

SUMMARY:
The study is a prospective registry. Consecutive patients with indications of implant / replacement or upgrade of pacemaker (PM), implantable cardioverter defibrillator (ICD), Implanted loop recorder (ILR) will be enrolled.

The primary objective of the study is to describe the clinical events during a long-term follow-up of non-selected population of patients implanted with an PM, ICD or ILR.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients underwent PM/ICD/ILR implantation
* Patient is willing and able to sign an authorization to use and disclose health information or an Informed Consent
* Patient must be able to attend all required follow-up visits at the study center for at least 12 months

Exclusion Criteria:

* No informed consent
* Patient is participating in another clinical study that may have an impact on the study endpoint

Exclusion Criteria:

* No informed consent

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study requires patients implanted with PM/ICD/ILR that meet all inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-01-07 (Actual); Primary Completion 2030-01-07 (Estimated); Study Completion 2050-01 (Estimated)

PRIMARY OUTCOMES:
CIEDs Infection | through study completion, an average of 1 year
  The number of patecipants with infections following implantation of cardiac implantable electronic devices
Appropriate ICD Therapies Antitachycardia pacing therapy or shock delivered by ICD for device detected ventricular arrhythmia | through study completion, an average of 1 year
  The number of partecipants with a least one episode of antitachycardia pacing therapy or shock delivered by ICD for device detected ventricular arrhythmias.
Inappropriate ICD Therapies | through study completion, an average of 1 year
  The number of partecipants with at least one episode of antitachycardia pacing therapy or shock delivered by ICD for device detected sopraventricular arrhythmias.

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Russo, MD PhD, Study Chair — University of Campania Luigi Vanvitelli
Locations (1):
- Vincenzo Russo, Naples, Napoli, Italy

IPD SHARING:
Plan to Share IPD: Undecided